CLINICAL TRIAL: NCT07252960
Title: Acute Effects of Warm Whirlpool Bath Therapy on Forearm and Hand Muscle Stiffness and Pain in Patients With Carpal Tunnel Syndrome: A Randomised Controlled Trial
Brief Title: Acute Effects of Warm Whirlpool Bath Therapy on Forearm and Hand Muscle Stiffness and Pain in Carpal Tunnel Syndrome
Acronym: CTS-WB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Collaborators: Amasya University (Other); Bangor University (Other)
Responsible Party: Principal Investigator, esedullah akaras, Dr., Erzurum Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETU-CTS-WB-2025-01
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal tunnel syndrome; Muscle stiffness; Whirlpool bath therapy
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Parallel-group randomized controlled trial with a 1:1 allocation ratio to warm whirlpool bath therapy or resting control.
Masking Description: Due to the nature of the intervention, neither participants nor treating therapists are blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm Whirlpool Bath Therapy (Experimental): Participants receive a single session of warm whirlpool bath therapy applied to the affected forearm and hand for 20 minutes.
  Interventions: Procedure: Warm Whirlpool Bath Therapy; Other: Resting Control Condition
- Resting Control (Active Comparator): Participants rest in a comfortable supported position for 20 minutes without whirlpool or thermal intervention.
  Interventions: Procedure: Warm Whirlpool Bath Therapy; Other: Resting Control Condition

INTERVENTIONS:
Procedure: Warm Whirlpool Bath Therapy — The affected hand and forearm are immersed in a therapeutic whirlpool bath with gently circulating water at approximately 38-39°C for 20 minutes. Participants are positioned to ensure comfort and muscle relaxation. Skin integrity and tolerance to heat are checked before treatment and monitored throughout the session
Other: Resting Control Condition — Participants rest in a comfortable supine or seated position with the affected forearm supported for 20 minutes. No active hydrotherapy, thermal or manual intervention is applied. Positioning and monitoring are comparable to the experimental group.

SUMMARY:
Carpal tunnel syndrome (CTS) is a common entrapment neuropathy that causes pain, paresthesia and functional limitations in the hand and wrist. Hydrotherapy methods such as warm whirlpool baths are frequently used in physiotherapy practice to reduce pain and improve soft-tissue properties, but their acute effects on forearm and hand muscle stiffness in CTS have not been clearly quantified.

This randomized controlled trial aims to investigate the acute effects of a single session of warm whirlpool bath therapy on forearm and hand muscle stiffness and pain intensity in adults with CTS. Participants diagnosed with CTS will be randomly allocated to an experimental group receiving a 20-minute warm whirlpool bath or to a resting control group. Muscle stiffness of selected forearm and hand muscles will be assessed using the MyotonPRO device, and pain intensity will be recorded with a numeric rating scale, immediately before and after the intervention. It is hypothesized that warm whirlpool bath therapy will produce a greater reduction in muscle stiffness and pain compared with rest alone.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is one of the most prevalent peripheral entrapment neuropathies and is characterized by pain, numbness and tingling in the hand, weakness of thenar muscles and impairments in hand function. In addition to nerve compression, changes in the mechanical properties of muscles and tendons surrounding the wrist and hand may contribute to symptoms, altered biomechanics and functional limitations in individuals with CTS. Increased muscle stiffness can restrict motion, impair force transmission and exacerbate pain, whereas excessive reductions in stiffness may compromise joint stability and fine motor control. Therefore, non-invasive interventions that can modulate muscle stiffness and relieve pain are of considerable interest in the management of CTS.

Warm whirlpool bath therapy is a traditional hydrotherapy modality that combines thermal and mild mechanical stimulation through circulating water. The convective heat may enhance local blood flow, reduce muscle spasm and alter viscoelastic properties of soft tissues, while water movement provides gentle massage-like effects. Although whirlpool baths are widely used in physiotherapy and rehabilitation practice, there is limited objective evidence regarding their acute effects on muscle mechanical properties in patients with CTS. Advances in handheld myotonometry devices, such as the MyotonPRO, allow non-invasive, reliable quantification of muscle stiffness, tone and elasticity and provide an opportunity to evaluate treatment effects beyond subjective palpation and self-reported outcomes.

This single-center, parallel-group randomized controlled trial will be conducted in a university physiotherapy and rehabilitation clinic. Physically active adults aged 18-65 years with a clinical diagnosis of carpal tunnel syndrome will be screened according to predefined inclusion and exclusion criteria. Eligible participants will be randomly assigned in a 1:1 ratio to either the warm whirlpool bath group or the resting control group. All assessments and interventions will be carried out on the affected upper limb.

In the experimental group, the affected hand and forearm will be immersed in a therapeutic whirlpool bath with gently circulating water at approximately 38-39°C for 20 minutes. Participants will be positioned to ensure comfort and muscle relaxation, and skin integrity and tolerance to heat will be monitored throughout the session. In the control group, participants will rest in a comparable position with the affected forearm supported for the same duration (20 minutes) without any active hydrotherapy or thermal intervention.

Outcome measures will be obtained immediately before and after the single intervention session. The primary outcomes are dynamic stiffness (N/m) of selected muscles of the forearm and hand (e.g., abductor pollicis brevis, flexor digitorum superficialis, extensor carpi radialis brevis, flexor carpi ulnaris) measured using the MyotonPRO device, and pain intensity at the wrist/hand assessed with a 0-10 numeric rating scale. Secondary outcomes may include additional MyotonPRO parameters such as muscle tone (frequency) and elasticity (logarithmic decrement). The main analysis will compare pre- to post-intervention changes between the whirlpool and control groups.

The overarching aim of this study is to provide objective, quantitative data on the acute effects of warm whirlpool bath therapy on muscle mechanical properties and pain in patients with CTS. Demonstrating a beneficial effect on muscle stiffness and pain may support the use of this simple, low-cost and non-pharmacological modality as part of comprehensive rehabilitation programs for carpal tunnel syndrome and inform future research on longer-term interventions and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Being apparently healthy without a known chronic systemic disease
* Physically active participants, regardless of gender
* Adults aged 18-65 years diagnosed with carpal tunnel syndrome
* No history of other chronic musculoskeletal or neurological disorders
* Not having any acute upper limb injury

Exclusion Criteria:

* Having a previous surgery on the affected wrist or hand
* Systemic conditions affecting nerve function, such as diabetes mellitus or thyroid disease
* Having a cardiovascular disease or uncontrolled hypertension
* Being younger than 18 or older than 65 years
* Being pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Primary | Baseline (pre-intervention) and immediately after the single 20-minute session (within approximately 5 minutes)
  Dynamic muscle stiffness (N/m) of selected muscles on the affected upper limb (abductor pollicis brevis, flexor digitorum superficialis, extensor carpi radialis brevis, flexor carpi ulnaris) measured with the MyotonPRO device. For each muscle, three consecutive measurements will be recorded and the mean value will be used for analysis. The primary outcome is the change in stiffness from baseline to post-intervention, compared between the warm whirlpool bath group and the resting control group. Higher values indicate greater muscle stiffness.

SECONDARY OUTCOMES:
Change in Pain Intensity in the Affected Hand/Wrist | Baseline (pre-intervention) and immediately after the single 20-minute session (within approximately 5 minutes)
  Patient-reported pain intensity at the affected hand/wrist assessed using a 0-10 numeric rating scale (0 = no pain, 10 = worst imaginable pain). The primary outcome is the change in pain score from baseline to post-intervention, compared between the warm whirlpool bath group and the resting control group. A decrease in score indicates pain reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan YAĞIZ, Principal Investigator — Amasya University
Locations (1):
- Erzurum Şehir Hastanesi, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. This is a single-center study with a relatively small sample size and a specific clinical population, which increases the risk of indirect re-identification even after de-identification. In addition, the current ethical approval and informed consent procedures do not explicitly cover external data sharing, and the study team has limited resources to support and monitor secondary data use. Aggregate results (e.g., group means and standard deviations) will be reported in scientific publications and presentations.